CLINICAL TRIAL: NCT03658902
Title: Retrospective Epidemiological Study on Patients Admitted for Botulism Poisoning in Intensive Care Units in France
Brief Title: Retrospective Epidemiological Study on Botulism in Intensive Care Units in France
Acronym: BotuREA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Other Study IDs: CHM-2017-538/05
Record Dates: First submitted 2018-08-31; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Botulism; Poisoning
Keywords: Botulism; Intensive Care
MeSH Terms: conditions — Botulism; Poisoning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Botulism poisoning is a rare but serious illness. Because of it's low incidence, it is not well known by physicians. Most studies describing botulism date back to the last century and do not take into account recent advances in intensive care.

The objective of this study is to describe the clinical course, interventions and outcomes of patients with severe botulism poisoning requiring a hospitalisation in an intensive care or high dependancy unit.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of botulism
* Admission in an intensive care or high dependancy unit

Exclusion Criteria:

* None

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients 15 years of age or older with a clinical diagnosis of botulism.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Survival | 2000 to 2017
  Proportion of patients alive at ICU discharge

SECONDARY OUTCOMES:
Age | 2000 to 2017
  Mean age of recruited patients
Weight | 2000 to 2017
  Mean weight of recruited patients
Height | 2000 to 2017
  Mean Height of recruited patients
History of motor impairment measured by the modified Rankin scale | 2000 to 2017
  History of neurological disorder with motor impairment before the poisoning, measured by the Modified Rankin Scale (0 to 6, 0 being no symptoms and 6 being deceased).
History of heart failure measured by the NYHA (New York Health Association) score | 2000 to 2017
  History of heart failure before the poisoning, measured by the NYHA (New York health Association) dyspnoea score (1 to 4, 1 being no symptoms and no limitation in daily physical activity, 4 being severe symptoms even at rest).
History of chronic respiratory failure: use of daily oxygen therapy AND/OR non invasive ventilation | 2000 to 2017
  Chronic respiratory failure defined by the use of chronic oxygen therapy AND/OR daily non invasive ventilation.
History of chronic kidney disease measured by the glomerular filtration rate. | 2000 to 2017
  History of chronic kidney disease before the poisoning, defined as a glomerular filtration rate < 60 mL/min/1.73m for more than 3 months OR chronic dialysis.
History of cirrhosis as measured by the CHILD-PUGH score. | 2000 to 2017
  Presence or absence of Cirrhosis, as measured by the CHILD-PUGH score (class A, B or C, A predicting a one year survival probability of 100%, C predicting a one year survival probability of 45%).
Source of the contamination | 2000 to 2017
  Suspected origin of the toxin: food poisoning, dermal wound, intravenous drug use, intestinal colonisation by Clostridium sp. or unknown.
Isolated or multiple cases | 2000 to 2017
  Whether the poisoning is isolated or one of multiple cases originating from the same source.
Botulinum Toxin type if identified | 2000 to 2017
  Botulinum toxin type if identified (A,B,C,D,E,F,G or H type toxin).
Severity at ICU admission | 2000 to 2017
  Simplified acute physiology score 2 (SAPS 2) at admission in the ICU: from 0 to 163, with 0 predicting a mortality risk of 0% and 163 of 100%.
Mechanical ventilation requirement | 2000 to 2017
  Whether the patient required or not mechanical ventilation during his ICU stay
Invasive mechanical ventilation requirement | 2000 to 2017
  Whether the patient required or not invasive mechanical ventilation during his ICU stay
Non invasive mechanical ventilation requirement | 2000 to 2017
  Whether the patient required or not non invasive mechanical ventilation during his ICU stay
Whether or not the patient required a tracheotomy during his ICU stay. | 2000 to 2017
  Whether the patient required a tracheotomy during his ICU stay
Enteral or parenteral nutritional support | 2000 to 2017
  Whether the patient required or not enteral or parenteral nutritional support during his ICU stay
Number of days of vasopressor support | 2000 to 2017
  Number of days the patient required vasopressor support during his ICU stay
Acute kidney injury measured by maximum serum creatinine during ICU stay. | 2000 to 2017
  Whether the patient developped an acute kidney injury during his ICU stay: measured by maximum serum creatinine during ICU stay in µmol/L.
Severe liver failure | 2000 to 2017
  Whether the patient developped an acute severe liver failure during his ICU stay, defined as a prothrombin time less than 50% due to liver failure.
Whether or not antitoxin was administered to the patient. | 2000 to 2017
  Whether botulinum antitoxin was administered.
Whether or not guanidine was administered during ICU stay | 2000 to 2017
  Whether guanidine was administered as a treatment for the botulinum poisoning.
Length of stay. | 2000 to 2017
  Number of hospitalisation days in the ICU.
Healthcare acquired infection | 2000 to 2017
  Whether the patient acquired a healthcare related infection during his stay in the ICU.
Mechanical ventilation related complications. | 2000 to 2017
  Whether the patient had any mechanical ventilation related complications during his stay in the ICU.
Bedrest complications: bedsores | 2000 to 2017
  Whether the patient acquired bedsores during his ICU stay.
Bedrest complications: thrombo-embolic complications | 2000 to 2017
  Whether the patient acquired thrombo-embolic complications (deep vein thrombosis or pulmonary embolism) during his ICU stay.
Disability at ICU discharge | 2000 to 2017
  Modified Rankin scale at ICU discharge, from 0 to 6, with 0 being asymptomatic and 6 being death.
Disability at hospital discharge | 2000 to 2017
  Modified Rankin scale at hospital discharge, from 0 to 6, with 0 being asymptomatic and 6 being death.
Last known disability | 2000 to 2017
  Last known modified Rankin scale, from 0 to 6, with 0 being asymptomatic and 6 being death.
Survival at hospital discharge | 2000 to 2017
  Proportion of patients alive at hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Guitton, MD, Principal Investigator — Centre Hospitalier le Mans